CLINICAL TRIAL: NCT00968266
Title: Improving Beliefs About Medication in Patients With Rheumatoid Arthritis: Randomized Controlled Study Into the Effect of a Motivational Patient-centered Intervention for Non-adherent Patients Compared to Usual Care Controls
Brief Title: Improving Beliefs About Medication in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sint Maartenskliniek (Other)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Joke Vriezekolk, Senior researcher, Sint Maartenskliniek
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RR-56-BMQ
Record Dates: First submitted 2009-08-27; First posted 2009-08-28 (Estimated); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Musculoskeletal Diseases; Rheumatoid Arthritis
Keywords: Adherence; Compliance; Rheumatoid Arthritis; Intervention; Beliefs about medication; Motivational Interviewing; Medication adherence; Patient compliance; Intervention studies
MeSH Terms: conditions — Musculoskeletal Diseases; Arthritis, Rheumatoid; Patient Compliance; Medication Adherence

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group intervention (Experimental): In short, the intervention consists of two group sessions moderated by a pharmacist. During these sessions, patients' self-perceived needs to take medication ('necessity beliefs'), concerns about taking medication ('concern beliefs'), and practical barriers are discussed. To explore a patient's individual ambivalence regarding his/her beliefs and barriers, the pharmacist uses Motivational Interviewing techniques. In between the sessions, participants make a homework assignment about their own beliefs and barriers, and eight weeks after the second session, a follow-up call to the individual patients is made by the pharmacist.
  Patients in the experimental arm also receive a brochure about the DMARDs they currently use (see: control arm)
  Interventions: Behavioral: Patient-centered group intervention
- Control arm: usual care (Active Comparator): In the control arm, patients receive a brochure about the DMARDs they are currently using.
  Interventions: Behavioral: Patient-centered group intervention

INTERVENTIONS:
Behavioral: Patient-centered group intervention — Session 1: Group discussion about the personal barriers for medication adherence. Supervisor: Pharmacist. Duration: 90 minutes. Goal: After this session the patient is aware of the benefits and barriers of adherence. The individual barriers to adherence (concerns and practical problems) and necessity beliefs about medication are identified and discussed.
  Session 2: Group based education on benefits of medication and discussing personal concerns about medication, practical barriers and beliefs about the necessity of medication. Supervisor: Pharmacist and rheumatologist. Duration: 90 minutes. Goal: Improving realistic beliefs about medication, stimulating an equal relationship between patient and health professional and motivating patients to be adherent.

SUMMARY:
The purpose of this study is to determine if a short motivational patient-centered intervention for non-adherent patients is more successful in improving beliefs about medication (and adherence) compared to a usual care control group of non-adherent patients.

DETAILED DESCRIPTION:
Disease Modifying Anti Rheumatic Drugs (DMARDs) reduce disease activity and radiological progression and improve long term functional outcome in patients with Rheumatoid Arthritis (RA). However, adherence is a prerequisite for a drug to be effective. A previous study showed that 33% of the RA-patients using DMARDs are non-adherent. Non-adherence can not be attributed to a single cause, but is the result of a complex and individual decision process. An intervention should not only consider practical barriers, such as forgetfulness, but also cognitive and other psychological variables that might impact medication adherence. Therefore, an intervention was developed focusing primarily on the non-adherent patient's individual beliefs and barriers to adherence.

The effectiveness of this intervention will be evaluated in a randomized clinical trial. Primary outcome measure is beliefs about medication assessed with the Beliefs about Medicines Questionnaire (BMQ). Additionally, adherence and adherence-related variables will be measured with questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* RA according to the 1986 ACR criteria for at least 1 year
* Prescription of anti-rheumatic medication (DMARDs)
* Non-adherent patients (Compliance Questionnaire Rheumatology)

Exclusion Criteria:

* Co-morbidity (physical or psychological) that unables patient to participate in the intervention
* Illiteracy
* Inability to communicate in Dutch
* Participation in other studies with significant burden

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-09; Primary Completion 2011-03 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Beliefs about medication, which is measured with Beliefs about Medicines Questionnaire (BMQ) | 3 weeks before first intervention session (T0), 2 weeks after first intervention session (T1), 6 months after first intervention session (T3), 12 months after first intervention session (T4)

SECONDARY OUTCOMES:
Adherence, measured with Compliance Questionnaire Rheumatology (CQR), Medication Adherence Report Scale (MARS) and refill rates | 3 weeks before first intervention session (T0), 2 weeks after first intervention session (T1), 6 months after first intervention session (T3), 12 months after first intervention session (T4)
Self-efficacy, measured with Arthritis Self Efficacy Scale | 3 weeks before first intervention session (T0), 2 weeks after first intervention session (T1), 6 months after first intervention session (T3), 12 months after first intervention session (T4)
Satisfaction with information about medication, measured with Satisfaction with Information about Medicines Scale (SIMS) | 3 weeks before first intervention session (T0), 2 weeks after first intervention session (T1), 6 months after first intervention session (T3), 12 months after first intervention session (T4)
Physical functioning, measured with Health Assessment Questionnaire (HAQ), Rheumatoid Arthritis Disease Activity Index (RADAI) and Visual Analogue Scale Pain (VAS Pain) | 3 weeks before first intervention session (T0), 2 weeks after first intervention session (T1), 6 months after first intervention session (T3), 12 months after first intervention session (T4)
Psychological functioning, measured with Hospital Anxiety and Depression Scale (HADS) and Illness Cognition Questionnaire (ICQ) | 3 weeks before first intervention session (T0), 2 weeks after first intervention session (T1), 6 months after first intervention session (T3), 12 months after first intervention session (T4)

CONTACTS AND LOCATIONS:
Overall Officials: Hanneke Zwikker, MSc, Principal Investigator — Sint Maartenskliniek; Bart van den Bemt, Principal Investigator — Sint Maartenskliniek
Locations (1):
- Sint Maartenskliniek, Nijmegen, Netherlands